CLINICAL TRIAL: NCT06171568
Title: Study of the One-year Outcomes of Patients Hospitalized in the Lariboisière Neurosurgery Department
Brief Title: Lariboisière Cognitive Assessment: Evaluation of the 1-year Outcomes
Acronym: ECOG
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: SBT Human(s) Matter (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP230528; 2023-A00386-39 (Other: IDRCB)
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Brain Injuries
Keywords: Brain injuries; Prognosis; Cognitive impairment; Cognition; Executive Function; Neuropsychological tests; Neuro-rehabilitation
MeSH Terms: conditions — Brain Injuries; Cognitive Dysfunction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tests and questionnaires — 1 year after discharge from neurosurgery department, included patients will answer to the:
  * Modified Rankin Scale;
  * Instrumental Activities of Daily Living (IADL) questionnaire;
  * Montreal Cognitive Assessment (MoCA);
  * Frontal assessment battery (BREF);
  * Rivermead questionnaire;
  * Short Form (36) Health Survey (SF-36)
  * Community Integration Questionnaire - Revised (CIQ-R)
  * Posttraumatic stress disorder CheckList (PCL-5)

SUMMARY:
Cognitive sequelae are common following acquired brain injuries. However, their detection can be challenging, particularly in acute care units such as neurosurgery. Specific screening in acute phase is critical for early detection and proper orientation. The Lariboisière cognitive assessment (Cog-First) is a brief cognitive evaluation conducted on a touch-screen tablet for patients with acquired brain injuries in the acute phase, which is integrated into routine care in Lariboisière.

The objective of this project is to evaluate the one-year cognitive and functional outcomes of patients who have undergone hospitalization in neuro-surgery. The primary aim is to assess whether the systematic pre-discharge assessment (Cog-First) performed as part of routine care can predict a poor functional prognosis and help identify at-risk patients earlier and more effectively.

DETAILED DESCRIPTION:
Traumatic brain injuries (TBI) are responsible for about 262 hospitalizations per 100,000 inhabitants in Europe each year. After a traumatic brain injury, 704 out of 100,000 individuals experience long-term consequences, including motor and/or balance disorders, fatigue, chronic pain, psychological disorders, and cognitive impairments such as memory problems, difficulties in comprehension, attentional deficits, and impairment of working memory. Without adequate rehabilitation, cognitive impairments can persist for several years, leading to significant socio-professional consequences such as job loss and social isolation, as well as medical and economic consequences.

The Paris TBI study showed that upon discharge from acute care services, only 45% of patients who had suffered severe traumatic brain injuries were referred to specialized rehabilitation facilities, while 30% returned directly home. Additionally, there is a lack of cognitive assessment in acute care services. For instance, in services that treat stroke patients, only 61% of patients will meet with a rehabilitation professional before their discharge. Short cognitive screening batteries typically used in the acute phase to guide patients' discharge from the hospital include the Montreal Cognitive Assessment (MoCA) or the Mini-Mental State Examination (MMSE). However, these scores are not very specific or sensitive, are examiner-dependent, and require trained personnel. Currently, there are few validated digital cognitive assessment batteries available for acute-phase evaluation and routine use in traumatic brain injury patients. Furthermore, evaluating cognitive impairments early after a traumatic brain injury can be challenging due to various confounding factors (e.g., fatigue, stressful hospitalization context) and organizational factors. Nevertheless, early assessment of cognitive impairments remains essential in order to appropriately refer patients, if necessary, to specialized rehabilitation facilities.

To address the need for better early detection of cognitive impairment following brain injuries, the investigators have developed the Cognitive Evaluation of Lariboisière (also known as Cog-First), a screening battery for cognitive impairments on a tablet device that can be quickly and independently completed by patients. Cog-First is now integrated into routine care in Lariboisière as a systematic pre-discharge assessment for patients discharged home without rehabilitation plan.

The main goal of this project is to identify patients who are at risk of experiencing cognitive impairments that could significantly impact their long-term functional prognosis. The investigators will evaluate whether the initial results obtained through the systematic evaluation using Cog-First at the time of discharge can accurately predict the functional and cognitive outcomes at one year. This could enable us to identify at-risk patients before discharge from acute care and refer them to specialized rehabilitation units earlier, leading to improved future outcomes for these individuals.

During the 1-year follow-up consultation after hospital discharge, eligible patients will be offered the opportunity to participate in the study. If they consent, their functional and cognitive abilities will be assessed using a set of tests and questionnaires. The assessments will include the modified Rankin score, IADL questionnaire, MoCA, Bref, Rivermead questionnaire, SF-36 questionnaire, CIQ-R questionnaire, and PCL-5 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient hospitalized in neurosurgery unit at Lariboisière hospital between February 2023 and February 2024
* Patient discharged home
* Patient affiliated to the social security system
* Patient having expressed no opposition

Exclusion Criteria:

* Patient transferred to a rehabilitation facility following hospitalization in neurosurgery
* History of neurological or psychiatric illness
* Severe uncorrected visual impairment and/or aphasia
* Non-French-speaking patients
* Patients receiving State Medical Aid (AME)
* Patients under guardianship/curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized at Lariboisière hospital in neurosurgery unit between February 2023 and February 2024.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the functional outcome at 1 year of patients who were hospitalized in the Lariboisière neurosurgery department compared with the initial systematic cognitive assessment (Cog-First) | 1 year
  The Modified Rankin Scale (MRS) will be used during the systematic follow-up consultation. The MRS is a score allowing functional independence level notation from 0 (no symptoms or incapacity) to 5 (severe disability).

SECONDARY OUTCOMES:
Assessment of the independence of patients in their daily life. | 1 year
  The Instrumental Activities of Daily Living (IADL) questionnaire will be submitted to patients.
  The IADL questionnaire gives a score going from 0 to 8. Higher score mean a better outcome.
Mesure of different cognitive functions of patients (language, memory, visio-spatial functions, attention, concentration, orientation in time and space). | 1 year
  Montreal Cognitive Assessment (MoCA) will be the used tool to answer this outcome.
  The MoCA gives a score going from 0 to 30. Higher score mean a better outcome.
Assess various cognitive functions in patients, including language, memory and visio-spatial abilities | 1 year
  The "Batterie Rapide d'Efficience Frontale" (BREF) test is a frontal assessment battery which will be used to question patients.
  The BREF test gives a score going from 0 to 18. Higher score mean a better outcome.
Rivermead questionnaire | 1 year after discharge from Neurosurgery department of Lariboisière
  Assessment of the post-concussion syndrome. The Rivermead questionnaire gives a score going from 0 to 52. Higher score mean a worse outcome.
Short Form (36) Health Survey (SF-36) | 1 year after discharge from Neurosurgery department of Lariboisière
  Assessment of quality of life. The SF-36 gives a score going from 0 to 100. Higher score mean a better outcome.
Community Integration Questionnaire - Revised (CIQ-R) | 1 year after discharge from Neurosurgery department of Lariboisière
  Assessment of socio-professional reintegration. The CIQ-R gives a score going from 0 to 35. Higher score mean a better outcome.
Posttraumatic stress disorder CheckList (PCL-5) | 1 year after discharge from Neurosurgery department of Lariboisière
  Assessment of post-traumatic stress. The PCL-5 gives a score going from 0 to 80. Higher score mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Mandonnet, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Alexis Schnitzler, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Neurosurgery - Lariboisière hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peeters W, van den Brande R, Polinder S, Brazinova A, Steyerberg EW, Lingsma HF, Maas AI. Epidemiology of traumatic brain injury in Europe. Acta Neurochir (Wien). 2015 Oct;157(10):1683-96. doi: 10.1007/s00701-015-2512-7. Epub 2015 Aug 14. PMID 26269030
- [Background] Jourdan C, Azouvi P, Genet F, Selly N, Josseran L, Schnitzler A. Disability and Health Consequences of Traumatic Brain Injury: National Prevalence. Am J Phys Med Rehabil. 2018 May;97(5):323-331. doi: 10.1097/PHM.0000000000000848. PMID 29016402
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Background] Stocchetti N, Zanier ER. Chronic impact of traumatic brain injury on outcome and quality of life: a narrative review. Crit Care. 2016 Jun 21;20(1):148. doi: 10.1186/s13054-016-1318-1. PMID 27323708
- [Background] Jourdan C, Bayen E, Bosserelle V, Azerad S, Genet F, Fermanian C, Aegerter P, Pradat-Diehl P, Weiss JJ, Azouvi P; Members of the Steering Committee of the PariS-TBI Study. Referral to rehabilitation after severe traumatic brain injury: results from the PariS-TBI Study. Neurorehabil Neural Repair. 2013 Jan;27(1):35-44. doi: 10.1177/1545968312440744. Epub 2012 Mar 28. PMID 22460612
- [Background] Schnitzler A, Erbault M, Solomiac A, Sainte Croix D, Fouchard A, May-Michelangeli L, Grenier C. Early rehabilitation after stroke: Strong recommendations but no achievement in the French Acute Healthcare Facilities. Ann Phys Rehabil Med. 2019 Jan;62(1):58-59. doi: 10.1016/j.rehab.2018.07.001. Epub 2018 Jul 19. No abstract available. PMID 30031892
- [Background] Rodrigues JC, Becker N, Beckenkamp CL, Mina CS, de Salles JF, Bandeira DR. Psychometric properties of cognitive screening for patients with cerebrovascular diseases A systematic review. Dement Neuropsychol. 2019 Jan-Mar;13(1):31-43. doi: 10.1590/1980-57642018dn13-010004. PMID 31073378
- [Background] de Guise E, Leblanc J, Champoux MC, Couturier C, Alturki AY, Lamoureux J, Desjardins M, Marcoux J, Maleki M, Feyz M. The mini-mental state examination and the Montreal Cognitive Assessment after traumatic brain injury: an early predictive study. Brain Inj. 2013;27(12):1428-34. doi: 10.3109/02699052.2013.835867. Epub 2013 Oct 8. PMID 24102622